CLINICAL TRIAL: NCT02946905
Title: Neurovascular Determinants of Cognitive Function in Adults With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Enrico M Novelli, Assistant Professor of Medicine, University of Pittsburgh
Other Study IDs: 12040139
Record Dates: First submitted 2016-09-26; First posted 2016-10-27 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — blood biomarkers of inflammation and oxidative damage
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SCD participant: No intervention
- Non-SCD participant: No intervention

SUMMARY:
Cognitive impairment is a poorly understood, serious, and emerging complication for adult patients with sickle cell disease. Because there is extensive microvascular damage from oxidative damage in sickle cell disease, the investigators hypothesize that this is also present in the cerebral microvasculature to cause cognitive impairment. The investigators plan to test this by correlating markers of inflammation and oxidative damage with cognitive performance and 7 Tesla brain MRI microvascular findings in these patients, with the long term goal of understanding the mechanisms and risk factors of cognitive impairment in sickle cell disease.

DETAILED DESCRIPTION:
The Neurovascular Determinants of Cognitive Function in Adults with Sickle Cell Disease is a study for adults 18 and older who have been diagnosed with Sickle Cell Disease (SCD). Many adult patients with SCD suffer from cognitive impairment (CI), a serious complication responsible for severe functional limitations, and whose pathogenesis, risk factors, and natural history are unknown. This research project will look at cognitive performance and 7 Tesla brain MRI findings along with markers of inflammation and oxidation to better understand the mechanism and risk factors. The investigators will complete a baseline assessment. SCD participants will be seen for follow-up at 3 and 5 years. Non-SCD participants will be seen for follow-up at 3 years. All assessments are completed at no cost and there is compensation for participation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above
2. Able to provide informed consent

For Non-SCD :

1. Between age 18 and 55
2. Able to provide informed consent
3. Are age, race, and gender matched to a Sickle Cell Disease study subject.

Exclusion Criteria:

1. Age less than 18 years
2. Current pregnancy or lactation
3. Any medical condition that may result in neurocognitive or brain dysfunction that is not secondary to SCD including:

   1. Diabetes mellitus
   2. Coronary artery disease
   3. Peripheral vascular disease
   4. Other causes of cerebral vasculitis such as Systemic Lupus Erythematosus (SLE)
4. Any contraindication to MRI scanning including:

   1. History of claustrophobia
   2. Presence of metallic implants such as cardiac pacemaker or implantable defibrillator, surgical aneurysm clips, or any implanted device (e.g. insulin pump, drug infusion device)
   3. Any known metal fragments embedded in the body (eg: ear implant)
   4. Neural stimulator (e.g. Transcutaneous Electrical Nerve Stimulation Unit)
   5. Metal in the eye (e.g. from machining)
   6. Any metallic foreign body, shrapnel, or bullet
   7. Inability to lie still for 30 minutes or more
5. Inability to provide direct consent
6. In a current medical or pain crisis as diagnosed by attending physician -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 150 participants with Sickle Cell Disease (SCD) 50 participants without Sickle Cell Disease
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2016-04; Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
7 Tesla MRI | 5 years
  Multiple conventional and novel markers of small vessel disease will be evaluated.

SECONDARY OUTCOMES:
Inflammation | 5 years
  Blood biomarkers of inflammation will be collected
Oxidative markers | 5 years
  Blood biomarkers of oxidative markers will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Novelli, MD, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No